CLINICAL TRIAL: NCT01601379
Title: Symptoms of Gastroesophageal Reflux Disease (GERD): Classification of Adult Subjects Suffering From Typical GERD Symptoms and Description of the Most Frequent Symptom Profiles and Characteristics - European Observational Study
Brief Title: Observational Study (This Means That no Drug is Tested) in Patients Suffering of Gastroesophageal Reflux Disease.
Acronym: PROFILE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016519; RABGRD4048 (Other: Janssen CTMS ID)
Record Dates: First submitted 2012-03-22; First posted 2012-05-18 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Gastroesophageal Reflux Disease; Gastro-oesophageal Reflux; Gastro-Esophageal Reflux; Esophageal Reflux; GERD
Keywords: Observational; GERD; Gastroesophageal Reflux Disease; Gastro-oesophageal Reflux; Heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study (this means that no drug is being tested in this study) is to obtain updated and detailed information about the Gastroesophageal Reflux Disease (GERD) specificities in European patients. The information about patients suffering from typical GERD symptoms will be collected in order to establish a classification of adult patients profile based on the characteristics of GERD symptoms. This study will only involve data collection about the disease. The treatment will not be affected by the study.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is one of the most common disorders seen by primary care providers and gastroenterologists in the United States and Europe. GERD is more than just heartburn, which is only one of several complaints. Patients can also suffer from regurgitation, nausea, sore throat, cough, hiccups, chest pain, sleep disturbance, etc. Individuals with the typical GERD symptoms (heartburn and/or acid regurgitation) constitute a diverse group. The detailed characterization of the different symptoms and their associations, but also their link with clinical or epidemiologic factors (age, body mass index [BMI], history of GERD, comorbidities, etc.), would help the physician to better individualize patient profiles and to adapt GERD management, enabling a better therapeutic response. In many studies the relationship between obesity and GERD has been looked at. However, the results of these studies are sometimes contradictory. The connection between obesity and elevated risk of GERD symptoms has been reported, although study results were sometimes contradictory (that is some of the studies showed that patients who were overweight did develop GERD symptoms more often than patients who had a normal weight; other studies did not show such a relationship). The purpose of this study is to update the data concerning adult patients suffering from GERD in European countries, as well as to explore the association between BMI and GERD symptoms, by determining the relative risks in patients belonging to different categories of BMI.This observational study will enroll patients who present at least 1 typical symptom of GERD (e.g., heartburn and/or regurgitation (the return of gastric content from the stomach to the mouth or throat)) in the week before inclusion in this study. The aim is to collect information about the symptom characteristics during one visit. During this visit, general information (age, weight, height,BMI), information about the medical history (including smoking and drinking habits, and drug use), information about any other diseases and lifestyle habits and detailed information about GERD (such as when it was fist diagnosed, how long the symptoms are present and when they occur, how they are treated) will be collected. A physical examination will be performed, consisting of a weight and height measurement, calculation of the body mass index (BMI), and a measurement of the waist. During the visit, the next steps for the GERD therapy (including changes in life style habits) will be discussed and this information will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an established diagnosis of GERD according to the investigator, or an occurrence of at least 1 typical GERD symptom (i.e., heartburn or regurgitation) at least once a week during the last 3 months.
* Patient has presented at least 1 typical GERD symptom (i.e., heartburn or regurgitation) in the week preceding the study visit.

Exclusion Criteria:

* Exclusively atypical digestive or non-digestive symptoms (e.g., epigastralgia, respiratory disturbances, thoracic manifestations, etc.)
* Current or recent (less than 1 year) history of gastric or duodenal ulcer
* History of surgery of the upper digestive tract
* Tumor of the superior digestive tract or ENT system;
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from GERD and presenting at least 1 of the typical GERD symptoms (i.e., heartburn and/or regurgitation), at least once a week, in the week prior to the first (and only) study visit are candidates for documentation in this study.
Sampling Method: Probability Sample
Enrollment: 7964 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Classification of adult patients suffering from typical GERD symptoms | Day 1
  The primary objective is to determine a classification of adult patients based on the presence or absence of 13 signs and symptoms characterizing GERD.

SECONDARY OUTCOMES:
Association with weight related variables | Day 1
  The association will be explored between weight related variables (e.g., BMI classes, waist circumference) and the found classification of patients.
Association with GERD related factors | Day 1
  The association will be explored between other GERD related factors (e.g., history of GERD, treatment) and the found classification of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV

REFERENCES:
- See also: Symptoms of gastroesophageal reflux disease (GERD): Classification of adult subjects suffering from typical GERD symptoms and description of the most frequent symptom profiles and characteristics - European observational study — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2358&filename=CR016519_CSR.pdf